CLINICAL TRIAL: NCT04941118
Title: Evaluation of the Effect of Dextrose Prolotherapy on Pain and Function in Women With Myofascial Pain Syndrome
Brief Title: Myofascial Pain Syndrome and Dextrose Prolotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Halil Ogut, Assistant Professor Doctor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MustafaKUPMR-MPS
Record Dates: First submitted 2021-06-15; First posted 2021-06-28 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Efficacy of Dextrose Prolotherapy in Myofascial Pain Syndrome
Keywords: Myofascial pain, dextrose prolotherapy, neck disability
MeSH Terms: interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): Only saline and local anesthetic (lidocaine)
  Interventions: Drug: Local anesthetic and saline injection to the myofascial trigger point
- Dextrose prolotherapy group (Active Comparator): Dextrose, saline and local anesthetic (lidocaine)
  Interventions: Drug: Injection of dextrose, local anesthetic and saline to the myofascial trigger point

INTERVENTIONS:
Drug: Injection of dextrose, local anesthetic and saline to the myofascial trigger point — An injection of 5 ml of 5% dextrose prolotherapy using 2.5 ml 10% dextrose, 1 ml 2% local anesthetic (lidocaine), 1.5 ml 0.9% saline will be administered to the active group from at least 10 trigger points.
  Arms: Dextrose prolotherapy group
Drug: Local anesthetic and saline injection to the myofascial trigger point — A total of 5 ml of solution created by using 4 ml of 0.9% saline and 1 ml of 2% local anesthetic (lidocaine) will be administered to the control group, with at least 10 trigger points.
  Arms: Control group

SUMMARY:
Myofascial pain syndrome is characterized by the presence of hypersensitive points called trigger points that cause pain, tenderness, spasm, stiffness, limitation of movement, weakness, taut band within the muscle, and pain reflected by pressing in a muscle group or a single muscle.

Prolotherapy is a regenerative treatment method in the treatment of chronic musculoskeletal pain, in which an irritating solution is injected, often hypertonic dextrose, into painful ligament and tendon attachments and adjacent joint spaces.

In this study, it was aimed to examine the effect of prolotherapy application on pain, neck range of motion and neck disability in women with myofascial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 60 women aged 20-50 years with a diagnosis of myofascial pain syndrome

Exclusion Criteria:

* Cervical radiculopathy, cervical degeneration, neck surgery or trauma in the last year, injection history for myofascial pain syndrome in the last 6 months, cognitive impairment and fibromyalgia, rheumatoid arthritis, hypothyroidism, diabetes mellitus

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | First month post-treatment
  0-10 cm visual scale (0: no pain, 10: most severe pain)
Neck Disability Index | First month post-treatment
  It measures the functional state of the neck by scoring between 0-5 points according to the severity of pain, consisting of 20 questions.
Neck joint range of motion measurement | First month post-treatment
  Active neck range of motion, which shows the movement of the neck in all directions, is evaluated by goniometric measurement.

SECONDARY OUTCOMES:
Side effects | Through study completion, an average of 6 month.
  Edema, ecchymosis, hematoma, allergic reaction, exacerbation of pain, systemic or distant side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Tayfur Ata Sökmen Faculty of Medicine, Hatay, Turkey (Türkiye)

REFERENCES:
- [Background] Farpour HR, Fereydooni F. Comparative effectiveness of intra-articular prolotherapy versus peri-articular prolotherapy on pain reduction and improving function in patients with knee osteoarthritis: A randomized clinical trial. Electron Physician. 2017 Nov 25;9(11):5663-5669. doi: 10.19082/5663. eCollection 2017 Nov. PMID 29403602
- [Background] Rabago D, Patterson JJ, Mundt M, Kijowski R, Grettie J, Segal NA, Zgierska A. Dextrose prolotherapy for knee osteoarthritis: a randomized controlled trial. Ann Fam Med. 2013 May-Jun;11(3):229-37. doi: 10.1370/afm.1504. PMID 23690322